CLINICAL TRIAL: NCT05500976
Title: Metabolomics INItiative: Effects of a MEDiterranean-amplified vs Habitual Western Diet on Biomarker Signatures, Cardiometabolic Health, and the Microbiome
Brief Title: Metabolomics Initiative: Mediterranean-amplified vs Habitual Western Diet on Food Signatures, Health, and Microbiome
Acronym: Mini-MED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry); Purdue University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 21-4563; R01DK113957 (NIH); 2070 (Other Grant/Funding Number: National Cattlemen's Beef Association)
Record Dates: First submitted 2022-08-03; First posted 2022-08-15 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Dietary Habits
Keywords: Mediterranean diet; Foodomics; Metabolomics; Food-specific signatures; Cardiometabolic health; Microbiome
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Participants will complete a 16-week randomized cross-over semi-controlled feeding study comparing two isocaloric dietary interventions. The two diets will be a Mediterranean-amplified habitual/Western (mini-MED) diet, containing 500 kcal/day from Mediterranean target foods (such as raspberries, avocado, red bell pepper, basil, walnuts, chickpeas, oats, salmon) and their habitual/Western (Western) diet,
  Participants will be randomized (1:1) to start one of the dietary interventions, with subsequent assignment to the other upon completion of the first. A permuted block randomization scheme using block size of 2 and stratification by sex will be utilized to ensure balance between intervention order and number of males and females in each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mini-Med (Experimental): Mediterranean-amplified habitual/Western (mini-MED) diet, containing 500 kcal/day from Mediterranean target foods (such as raspberries, avocado, red bell pepper, basil, walnuts, chickpeas, oats, salmon).
  Interventions: Other: Semi-controlled dietary intervention - MiniMed
- Western (Active Comparator): Habitual/Western (Western) diet, containing 500 kcal/day from non-Mediterranean target foods (such as potato, beef, sour cream, refined grain bread, chocolate dessert).
  Interventions: Other: Semi-controlled dietary intervention - Western

INTERVENTIONS:
Other: Semi-controlled dietary intervention - Western — Participants will complete a 2-week washout prior to a 16-week randomized, crossover semi-controlled feeding study of mini-MED vs Western diet. Each diet intervention will last four weeks, with 500 kcal/day of target Western diet foods (eg, beef, potatoes, bread, sour cream) provided during each intervention and will be repeated twice.
  Arms: Western
Other: Semi-controlled dietary intervention - MiniMed — Participants will complete a 2-week washout prior to a 16-week randomized, crossover semi-controlled feeding study of mini-MED vs Western diet. Each diet intervention will last four weeks, with 500 kcal/day of target Mediterranean foods (eg, oatmeal, salmon, nuts, basil, olive oil, fruits) provided during each intervention and will be repeated twice.
  Arms: mini-Med

SUMMARY:
This study plans to learn more about how consuming a diet with foods typical to a Mediterranean Diet such as whole grains, fruits and vegetables in a Western-style diet compares to eating a typical Western-style diet. This study will look at how diet affects overall health including risk factors for heart disease, gut health and inflammation as well as underlying mechanisms linking whole food to health. Findings from this study will potentially inform effective dietary recommendations and interventions, thereby reducing chronic disease in humans.

DETAILED DESCRIPTION:
The investigators propose to conduct a 16-week randomized, cross-over, semi-controlled feeding study of two isocaloric dietary interventions: 1. Mediterranean-amplified habitual/Western (mini-MED) diet, containing 500 kcal/day from Mediterranean target foods (such as raspberries, avocado, red bell pepper, basil, walnuts, chickpeas, oats, salmon); and 2. Habitual/Western (Western) diet, containing 500 kcal/day from non-Mediterranean target foods (such as potato, beef, sour cream, refined grain bread, chocolate dessert); among individuals who are not already consuming a Mediterranean-style dietary pattern. Participants will have overweight or obesity and meet criteria for Metabolic Syndrome (MetS), and therefore be at increased risk of cardiometabolic disease (CMD).

The primary goal is to validate results from metabolomics analyses of foods and biospecimens from a completed Mediterranean-style dietary intervention in a prospective feeding trial. Secondary aims are to evaluate impacts of incremental changes in diet on cardiometabolic health and microbiome structure/function. The primary hypothesis is that pre-defined metabolomics signatures in participant biospecimens will be responsive to dietary intakes and reproducible within individuals over time. The secondary hypotheses are that a Mediterranean-amplified diet will lead to improvements in cardiometabolic health and changes in microbiome structure/function over time and compared to a habitual Western diet.

Aim 1: Test reproducibility of pre-defined signatures from Mediterranean target foods provided in mini-MED in biospecimens (blood/urine) within individuals over time. Participants will complete a 16-week randomized cross-over dietary intervention of mini-MED vs Western diet. The investigators hypothesize that: (1) novel food-specific compounds will increase in participant biospecimens after consumption of mini-MED and decrease during Western diet, and (2) established biomarkers of fruit/vegetable intake (e.g., plasma and skin carotenoids, urine polyphenols) and other target foods (e.g., plasma alkylresorcinols, astaxanthin) will increase after consumption of mini-MED.

Aim 2: Determine the impact of mini-MED on cardiometabolic health. Cardiometabolic health indicators (e.g., blood pressure, lipid panel, inflammatory cytokines, indicators of subclinical inflammation) will be assessed pre- and post- each intervention. The investigators hypothesize that consumption of mini-MED will lead to improvements in cardiometabolic health indicators (e.g., reductions in blood pressure, total cholesterol, LDL cholesterol, triglycerides, C-reactive protein, bioactive lipids; increases in HDL cholesterol) over time and compared to Western diet.

Aim 3: Evaluate changes in microbiota community structure/function in response to mini-MED. Microbiome structure (taxonomy) and function (metagenomics) will be assessed pre- and post- each intervention. The investigators hypothesize that consumption of mini-MED will lead to increases in microbiome diversity and enrichment in taxa associated with increased production of health-promoting compounds (e.g., short chain fatty acids) over time and compared to Western diet.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI 25-37 kg/m2) and weight-stable;
* Age 30-69 years;
* Nonsmoker (including tobacco, marijuana, and other inhaled substances);
* Consistent physical activity levels for 3 months prior to and throughout the study period;
* Stable medication use for 6 months prior to and throughout the study period;
* Having at least three components of Metabolic Syndrome (MetS): i.e., impaired fasting glucose, hypertension, central adiposity (waist circumference ≥ 94 cm or 80 cm, for men and women, respectively), fasting hypertriglyceridemia, and/or low levels of HDL cholesterol17 OR on medication for the treatment of hyperglycemia, hypertension, or hypercholesterolemia in lieu of meeting the corresponding MetS component;
* Report of baseline consumption of a habitual diet not meeting criteria for a Mediterranean-style dietary pattern, defined as a score of <5 as assessed via the Mediterranean Diet Assessment Tool
* Follows an omnivorous diet and willing to consume all provided foods (e.g., will eat salmon, fruits/vegetables, beef);
* Willingness to refrain from consumption of nutritional supplements, herbal supplements, botanical supplements, and pre- or probiotics aside from those prescribed by a physician for the duration of the study;
* Willingness to come to the CTRC biweekly for clinical assessments and biospecimen collection;
* No plans to relocate or for extended travel (>1 week) within next 6 months; and
* Capable and willing to provide informed consent

Exclusion Criteria:

* Use of medications contraindicating increased consumption of fruits/vegetables (e.g., warfarin);
* Diagnosis of acute or chronic condition impacting appetite, food intake, and/or the metabolism and absorption of foods to be provided (e.g., Crohn's disease, Celiac disease, Ulcerative colitis, short bowel syndrome, chronic diarrhea);
* Impaired liver or kidney function;
* Food allergies to foods provided in either dietary intervention;
* Vegetarian, vegan; and
* For females: pregnant or lactating or planning to become pregnant during study period

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Foodomics | Baseline to endline changes in food-specific compounds over each 4-week dietary intervention period
  Change in the number of unique to food compounds (i.e., putative biomarkers of intake) from baseline to end of each diet intervention period in participant serum samples.

SECONDARY OUTCOMES:
Cardiometabolic Health - IL-6 | Baseline to endline changes over each 4-week dietary intervention period
  Changes in blood inflammatory markers including IL-6 over time and between the two dietary interventions.
Cardiometabolic Health - TNF-alpha | Baseline to endline changes over each 4-week dietary intervention period
  Changes in blood inflammatory markers including TNF-alpha over time and between the two dietary interventions.
Cardiometabolic Health - C-reactive protein | Baseline to endline changes over each 4-week dietary intervention period
  Changes in blood inflammatory markers including C-reactive protein over time and between the two dietary interventions.
Cardiometabolic Health - alpha-1-acid glycoprotein | Baseline to endline changes over each 4-week dietary intervention period
  Changes in blood inflammatory markers including alpha-1-acid glycoprotein over time and between the two dietary interventions.
Cardiometabolic Health - Total Cholesterol | Baseline to endline changes over each 4-week dietary intervention period
  Changes in fasting total cholesterol over time and between the two dietary interventions.
Cardiometabolic Health - LDL Cholesterol | Baseline to endline changes over each 4-week dietary intervention period
  Changes in fasting LDL cholesterol over time and between the two dietary interventions.
Cardiometabolic Health - HDL Cholesterol | Baseline to endline changes over each 4-week dietary intervention period
  Changes in fasting HDL cholesterol over time and between the two dietary interventions.
Cardiometabolic Health - Triglycerides | Baseline to endline changes over each 4-week dietary intervention period
  Changes in fasting triglycerides over time and between the two dietary interventions.
Cardiometabolic Health - Blood Pressure | Baseline to endline changes over each 4-week dietary intervention period
  Changes in blood pressure over time and between the two dietary interventions.
Cardiometabolic Health - Insulin | Baseline to endline changes over each 4-week dietary intervention period
  Changes in fasting blood insulin over time and between the two dietary interventions.
Cardiometabolic Health - Glucose | Baseline to endline changes over each 4-week dietary intervention period
  Changes in fasting blood glucose over time and between the two dietary interventions.
Cardiometabolic Health - Adipokines | Baseline to endline changes over each 4-week dietary intervention period
  Changes in circulating plasma adipokines over time and between the two dietary interventions.
Gut Microbiota | Baseline to endline changes over each 4-week dietary intervention period
  Changes in diversity and community composition of the gut microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy F Krebs, MD, Principal Investigator — University of Colorado School of Medicine; Nichole Reisdorph, PhD, Principal Investigator — University of Colorado School of Pharmacy; Wayne Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
1) Data will be made available in accordance with the "Final NIH Statement on Sharing Research Data". Results, data, workflows, and tools will be made available through publication, presentations at scientific meetings, open access on our website following publication, in open repositories when they are established, and according to other policies set forth by the NIH. The primary type of data collected will be raw mass spectrometry data. There are widely available free-ware data converters for mass spectrometry data that have been created by the mass spectrometry community. Thus, the data from this project will be saved in the original raw format.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available within 12 months of publication of results for a minimum period of 3 years.

REFERENCES:
- [Derived] Hill EB, Tang M, Long JM, Kemp JF, Westcott JL, Hendricks AE, Reisdorph NA, Campbell WW, Krebs NF; mini-MED Trial Team. mini-MED: study protocol for a randomized, multi-intervention, semi-controlled feeding trial of a Mediterranean-amplified vs. habitual Western dietary pattern for the evaluation of food-specific compounds and cardiometabolic health. Trials. 2024 Feb 2;25(1):101. doi: 10.1186/s13063-024-07939-8. PMID 38302990
- [Derived] Hill EB, Reisdorph RM, Rasolofomanana-Rajery S, Michel C, Khajeh-Sharafabadi M, Doenges KA, Weaver N, Quinn K, Sutliff AK, Tang M, Borengasser SJ, Frank DN, O'Connor LE, Campbell WW, Krebs NF, Hendricks AE, Reisdorph NA. Salmon Food-Specific Compounds and Their Metabolites Increase in Human Plasma and Are Associated with Cardiometabolic Health Indicators Following a Mediterranean-Style Diet Intervention. J Nutr. 2024 Jan;154(1):26-40. doi: 10.1016/j.tjnut.2023.10.024. Epub 2023 Oct 31. PMID 37918675